CLINICAL TRIAL: NCT03078803
Title: A Prospective Multicenter Randomized Controlled Trial Comparing Fecal Microbiota Transplantation (FMT) to Placebo in the Treatment of Mild to Moderate Crohn's Disease
Brief Title: Fecal Transplant for Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: University of Calgary (Other); McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 66218
Record Dates: First submitted 2017-01-12; First posted 2017-03-13 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Crohn Disease
Keywords: fecal transplant; inflammatory bowel disease
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fecal microbiota transplant (Experimental): Transfer of healthy human gut bacteria
  Interventions: Biological: Fecal Microbiota Transplant (FMT)
- Placebo (Placebo Comparator): Water
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Fecal Microbiota Transplant (FMT) — FMT delivered by colonoscopy and oral capsules
  Other Names: FMT
  Arms: Fecal microbiota transplant
Biological: Placebo — Transfer of water only
  Arms: Placebo

SUMMARY:
To determine the efficacy and safety of serial FMT at inducing and maintaining clinical and endoscopic response in patients with mild to moderate Crohn's disease

DETAILED DESCRIPTION:
Double blind study will randomize patients with mild to moderate Crohn's 1:1 (FMT : water) stratified by disease duration and current use of biologic therapy. First FMT/placebo at week 0 by colonoscopy plus weekly FMT/placebo by capsules for 7 weeks. At week 8, a repeat colonoscopy will be done and endoscopy score repeated.

Responders in FMT arm are eligible to enter open label phase to receive FMT by capsules q2 weeks.

Blood, stool and urine samples, colonic biopsies will be collected. Quality of Life as measured by Short Inflammatory Bowel Disease Questionnaire, EuroQol five dimensions, and Work Productivity and Activity Impairment Questionnaire: Crohns disease and dietary intake diary collected.

Colonoscopies recorded and reviewed by a central reader.

ELIGIBILITY:
Inclusion Criteria:

* mild to moderate ileal, ileo-colonic or colonic Crohns disease
* active ileal and/or colonic disease on endoscopy with or without elevated inflammatory markers i.e. C-reactive protein >8mg/L, elevated fecal calprotectin >250 ug/g
* If applicable, meds stable as follows: 5-ASA for 4 weeks, prednisone up to 20mg QD for 4 weeks, budesonide up to 6mg QD for 4 weeks, azathioprine, 6-MP and methotrexate for 12 weeks
* Use of effective contraception

Exclusion Criteria:

* Antibiotic exposure within 30 days and probiotic exposure within 14 days
* topical inflammatory bowel disease therapy within 2 weeks
* active perianal disease
* requirement for concurrent antibiotic therapy
* SES-CD score <5
* severe CD HBI >25 or need for hospitalization
* abdominal abscess
* extensive colonic resection, subtotal or total colectomy
* ileostomy, colostomy, known fixed symptomatic stenosis or complex fistulae
* evidence of or treatment for C. difficile or other intestinal pathogen including Cytomegalovirus within 28 days
* requiring or expected to require surgical intervention
* history or evidence of adenomatous colonic polyps not removed
* history of evidence of colonic dysplasia
* active substance abuse or psychiatric problems that may interfere with study
* chronic Hep B, C, or HIV infection
* pregnancy or planning to become pregnant
* upper CD
* history of adhesions preventing colonoscopy to cecum
* planned bowel resection within 3 mon of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2022-08-29 (Actual)

PRIMARY OUTCOMES:
Clinical and Endoscopic Remission | Week 8
  Harvey Bradshaw Index <5 and Simple endoscopic score <5

SECONDARY OUTCOMES:
Clinical response | Week 8
  Harvey Bradshaw Index reduction by 3 points
Clinical remission | Week 8
  Harvey Bradshaw Index <5
Endoscopic response | Week 8
  Simple endoscopic score reduction by 50%
Endoscopic remission | Week 8
  Simple endoscopic score <5
Quality of Life 1 | Week 8
  Mean changes in Short Inflammatory Bowel Disease Questionnaire
Quality of Life 2 | Week 8
  Mean changes in Euro five dimensions questionnaire
Quality of Life 3 | Week 8
  Mean changes in Work Productivity and Activity Impairment: Crohns Disease questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Dina Kao, MD, Principal Investigator — University of Alberta
Locations (3):
- Canada (3):
  - Foothills Hospital, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - McMaster University, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kao D, Wong K, Jijon H, Moayyedi P, Franz R, McDougall C, Hotte N, Panaccione R, Semlacher E, Kroeker KI, Peerani F, MacDonald KV, Xu H, Narula N, Turbide C, Marshall DA, Madsen KL. Preliminary Results From a Multicenter, Randomized Trial Using Fecal Microbiota Transplantation to Induce Remission in Patients With Mild-to-Moderate Crohn's Disease. Am J Gastroenterol. 2024 Nov 12;120(6):1334-1344. doi: 10.14309/ajg.0000000000003196. PMID 39530534